CLINICAL TRIAL: NCT00990626
Title: Seroquel XR in Schizophrenia Relapse Prevention
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-NHU-SER-2009/1
Record Dates: First submitted 2009-10-01; First posted 2009-10-07 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Schizophrenia Relapse Prevention
Keywords: Seroquel XR; schizophrenia relapse prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Schizophrenic outpatients

SUMMARY:
The purpose of the study is to determine whether the Seroquel XR treatment for 6 months improve the relapse prevention in schizophrenic outpatients

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenic outpatients on at least 600 mg Seroquel XR treatment for at least 1 month

Exclusion Criteria:

* Severe cerebro- and cardiovascular disease, severe hepatic impairment, gravidity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Rate of patients remained relapse free after 6 months of treatment

SECONDARY OUTCOMES:
Adherence rate of patients
Quality of Life (QoL )

CONTACTS AND LOCATIONS:
Overall Officials: Attila Németh, Principal Investigator — National Psychiatric Centre; Lilla Szabó, Study Chair — AstraZeneca Hungary MC; Tamás Bábel, Study Director — AstraZeneca Hungary MC
Locations (48):
- Hungary (48):
  - Research Site, Baja
  - Research Site, Barcs
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Debrecen
  - Research Site, Dombóvár
  - Research Site, Dunaújváros
  - Research Site, Eger
  - Research Site, Egerszalók
  - Research Site, Emőd
  - Research Site, Esztergom
  - Research Site, Érd
  - Research Site, Gödöllő
  - Research Site, Gyöngyös
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Heves
  - Research Site, Hódmezővásárhely
  - Research Site, Jánoshalma
  - Research Site, Jászberény
  - Research Site, Kalocsa
  - Research Site, Kecskemét
  - Research Site, Kétegyháza
  - Research Site, Kiskunhalas
  - Research Site, Kistokaj
  - Research Site, Miskolc
  - Research Site, Nagyatád
  - Research Site, Nagykanizsa
  - Research Site, Nagykálló
  - Research Site, Nagykőrös
  - Research Site, Orosháza
  - Research Site, Pécs
  - Research Site, Pomáz
  - Research Site, Sátoraljaújhely
  - Research Site, Soltvadkert
  - Research Site, Sopron
  - Research Site, Sümeg
  - Research Site, Szeged
  - Research Site, Szeghalom
  - Research Site, Szekszárd
  - Research Site, Szentes
  - Research Site, Székesfehérvár
  - Research Site, Szigetszentmiklós
  - Research Site, Szigetvár
  - Research Site, Szolnok
  - Research Site, Szombathely
  - Research Site, Tatabánya
  - Research Site, Veszprém